CLINICAL TRIAL: NCT06416046
Title: Efficacy of Photobiomodulation in the Treatment and Relief of Pain in Recurrent Aphthous Stomatitis: a Randomized, Triple-blind, Controlled Clinical Trial
Brief Title: Efficacy of Photobiomodulation in the Treatment and Relief of Pain in Recurrent Aphthous Stomatitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Manoela Domingues Martins, Principal Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PMB and RAS
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Photobiomodulation; Stomatitis, Aphthous
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Intervention Model Description: Participants will be allocated and randomized into 2 groups: Group I: PBM (n=17) photobiomodulation intra oral high potency laser (4.5J) and Group II: control (n=17).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, examiner and outcomes assessor will not know which group has been allocated (triple-blind). Another person (the applicator) will carry out the randomization and know which group the patient belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intraoral photobiomodulation (PBM) (Experimental): A gallium-aluminum arsenide diode laser (Gemini® manufactured by Azena Medical, LLC, distributed by Ultradent Products, Inc.) with double wavelength 810 + 980 nm. The equipment will be programmed with 0,3W of power. The application of PBM will be carried out for at least 03 alternate days within 01 week by a trained professional. Patients who still have an ulcerated lesion on the 7th day will be assessed every 2 days until complete healing. During each irradiation, the applicator and patients will wear specific protective goggles and the instruments will be disinfected with an antiseptic solution (Chlorhexidine 2%).
  Points of application:
  Equidistant points (0.5cm) along the length of the lesion and in contact with the lesion.
  Interventions: Device: Gemini laser
- Placebo (Placebo Comparator): The application of placebo will be carried out for at least 03 alternate days within 01 week (3x within 07 days) by a trained professional. Patients who still have an ulcerated lesion on the 7th day will be assessed every 2 days until complete healing. The device will not be activated and the applicator and patients will wear specific protective goggles and the instruments will be disinfected with antiseptic solution (Chlorhexidine 2%).
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Gemini laser — Photobiomodulation (810 + 980 nm, 15s/point, 11.8J/cm²) to evaluate healing and pain relief in recurrent aphthous stomatitis. A 0.7mm intraoral tip will be used - spot 0.38cm2 on the extent of the lesion.
  Arms: Intraoral photobiomodulation (PBM)
Other: Placebo — Examination and follow-up until the lesion heals spontaneously. The laser will not be activated.
  Arms: Placebo

SUMMARY:
Photobiomodulation (PBM) is a therapy that stimulates repair, pain relief, and reduces inflammation. The aim of this study is to evaluate the effectiveness of a new PBM protocol in the treatment and pain relief of RAS lesions.

DETAILED DESCRIPTION:
Recurrent aphthous stomatitis (RAS) is the most common chronic ulcerative inflammatory disorder of the oral cavity, affecting approximately 20% of the general population, with no gender predilection. Its etiopathogenesis remains undefined, although factors such as local trauma and syndromes like Behcet's syndrome are implicated in predisposition. RAS manifests in three distinct clinical presentations, with the smallest being the most common, accounting for 80% of cases. Minor RAS present as round or oval ulcers, smaller than 1 cm, covered by a grayish-white pseudomembrane, commonly occurring on non-keratinized mucosa such as lips, buccal mucosa, and floor of the mouth. Photobiomodulation (PBM) is a therapy that stimulates repair, pain relief, and reduces inflammation. The aim of this study is to evaluate the effectiveness of a new PBM protocol in the treatment and pain relief of RAS lesions. The study is a randomized, triple-blind, placebo-controlled clinical trial to be conducted at the Hospital de Clinicas de Porto Alegre (HCPA) in Rio Grande do Sul, from March 2023 to December 2025. Thirty-four patients of both genders will be selected and randomly allocated into three groups: 17 patients in the PBM treatment group with 4.5J and 17 patients in the control group. Inclusion criteria are patients over 18 years old with at least one painful ulcer in the mouth. If the patient has more than one ulcer, all will be treated. Exclusion criteria include patients who have undergone previous treatment for RAS, patients with asymptomatic ulcers, and patients with any systemic condition related to RAS - for example, Behçet's Syndrome, Periodic Fever Syndrome, Aphthous Stomatitis, Pharyngitis, and Cervical Adenitis, HIV infection. The study outcome is lesion healing, and the independent variables analyzed in the study will be: pain, lesion size, and difficulty in eating, drinking, and brushing teeth due to the presence of RAS. These variables will be collected through questionnaires administered during all patient visits. Analyses will be performed using PASW 18.0 software. Initially, data distribution will be assessed using Shapiro-Wilk and Kolmogorov-Smirnov tests. If the data show normal distribution (p>0.05), the t-test will be used. If the distribution is non-normal (p<0.05), the Wilcoxon test will be employed. The significance level (p-value) will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients presenting at least one painful mouth ulcer (minor ulcer), located on the tongue, jugal mucosa or labial mucosa, starting on the same day or the day before.

Exclusion Criteria:

* Patients who have already undergone other treatment for RAS;
* Patients with asymptomatic ulcers;
* Patient must not be undergoing or have undergone any treatment for RAS;
* Patients with any systemic condition related to RAS - e.g. Behcet's Syndrome, Periodic Fever Syndrome, Pharyngitis and Cervical Adenitis, HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 1 week
  Pain will be assessed at all appointments using the Visual Analog Scale (VAS), which will be represented by a 10 cm straight line, where 0 corresponds to the best situation and 10 to the worst situation. The research subjects will be instructed by the evaluator to mark a point on the 10 cm line.
Assessment of ulcer size | 1 week
  Ulcer size will be assessed at every appointment using the tip of a millimeter-sized periodontal probe.
Functional assessment | 1 week
  The functional assessment will be carried out at all appointments, evaluating the patient's subjective experience of difficulty in eating, drinking and brushing their teeth due to the presence of RAS. The answers will be scored from 0 (no difficulty) to 4 (a lot of difficulty) according to the questionnaire given to the patients

SECONDARY OUTCOMES:
Time measurement | 1 week
  The time of all the sessions carried out will be timed with the aid of a stopwatch, starting at the beginning of the device's activation until its deactivation. The time in seconds will be recorded on the daily evaluation form.
Saliva collection | 1 week
  Saliva samples will be collected from participants at two clinical assessment points. Patients must abstain from eating or drinking for 30 minutes prior. Saliva is collected unstimulated, with patients seated, eyes open, head slightly tilted down, and refraining from speaking, swallowing, or mouth opening for 5 minutes. Samples are collected in sterile Falcon tubes, immediately placed on ice, and stored at -80°C for later inflammatory marker analysis. Samples are stored in HCPA's Biobank per regulations and analyzed at CPE, then discarded post-analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Manoela Martins, PhD, Study Director — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After publication of the outcomes, for one year
Access Criteria: If formally requested and referenced by the interested researcher